CLINICAL TRIAL: NCT04212754
Title: Management and Outcomes Following Emergency Surgery for Traumatic Brain Injury - a Multi-centre, International, Prospective Cohort Study (the Global Neurotrauma Outcomes Study)
Brief Title: Management and Outcomes Following Emergency Surgery for Traumatic Brain Injury
Acronym: GNOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, David Clark, Clinical Research Fellow in Global Neurotrauma, University of Cambridge
Other Study IDs: GNOS1
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Traumatic Brain Injury; Head Injury; Brain Injuries; Brain Trauma; Brain Injuries, Traumatic; Head Injury Trauma
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Procedure: Emergency surgery for traumatic brain injury
  Interventions: Other: Exposure: human development index of country

INTERVENTIONS:
Other: Exposure: human development index of country — Primary comparison: Between country groups defined by human development index.

SUMMARY:
Primary aim:

The primary aim of the study is to compare survival to discharge (or survival to 14 days post-operatively, whichever comes first) following emergency surgery for traumatic brain injury (TBI) across Human Development Index settings.

Primary outcome measure:

The primary outcome measure will be survival to discharge (or survival to 14 days post-operatively, whichever comes first)

Primary comparison:

Between country groups defined by human development index.

Centre eligibility:

Any hospital or clinic worldwide performing emergency surgery for traumatic brain injury is eligible to participate.

Patient eligibility:

All adult and paediatric patients admitted to the participating institution with a traumatic brain injury for which they receive emergency surgery during the selected 30-day inclusion period are eligible for inclusion in the study.

Team:

Individual hospital teams with up to four people, collecting data for 30 days.

Time period:

Local study teams may select any 30-day period from the 1st of November 2018 and the 31st of December 2019 to start their study. Patients operated on who meet the inclusion criteria between 00:01 on day 0 and 23:59 on day 30 of the selected study period will be included.

Validation:

We will employ a method of data validation in every centre that will give us a quantitative estimate of case ascertainment that is feasible even in low-resource centres.

ELIGIBILITY:
Centre Inclusion Criteria:

Any hospital or clinic worldwide performing emergency surgery for traumatic brain injury is eligible to participate. In the majority of institutions, emergency surgery for TBI is provided by neurosurgeons - however, centres in which emergency surgery for TBI is provided general surgeons, trauma surgeons, general medical doctors or even non-physician clinicians are also eligible to participate.

Inclusion Criteria:

- All adult and paediatric patients admitted to the participating institution with a traumatic brain injury for which they receive emergency surgery during the selected 30-day inclusion period are eligible for inclusion in the study.

Exclusion Criteria:

* Patients who only have an external ventricular drain or intraparenchymal wire (or other monitoring device) inserted for the diagnosis and/or management of intracranial hypertension.
* Patients who undergo procedures for chronic subdural haematoma(s), including burr holes or mini-craniotomies.
* Elective (planned admission) or semi-elective (where patient initially admitted as an emergency, then discharged from hospital, and re-admitted at later time for surgery) procedures.
* Patients who have previously had emergency cranial surgery for traumatic brain injury rendering them eligible for inclusion in this study (regardless of whether they were included)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients undergoing emergency surgery for traumatic brain injury.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-02-13 (Estimated); Study Completion 2020-02-29 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality (or 14 day mortality, whichever comes first) | Up until hospital discharge, death or 14 days postoperatively, whichever comes first

SECONDARY OUTCOMES:
Perioperative complications: Return to operating theatre | Up until hospital discharge, death or 14 days postoperatively, whichever comes first
  Including reason for return.
Perioperative complications: Surgical site infection (SSI) | Up until hospital discharge, death or 14 days postoperatively, whichever comes first
  SSI is stratified into superficial and deep/organ space infection.
Length of stay in hospital (days) | Up until hospital discharge, death or 14 days postoperatively, whichever comes first
Length of stay in intensive care (days) | Up until hospital discharge, death or 14 days postoperatively, whichever comes first
  For patients admitted to intensive care.
Glasgow Coma Score at discharge/end of follow up period | At hospital discharge 14 days postoperatively, whichever comes first
  3-15, 3 signifies no eye opening, verbal response or motor response to painful stimulus, 15 signifies no impairment to consciousness. For patients surviving to discharge and/or 14 days postoperatively.
Location that the patient was discharged to | Within 14 days post-operatively, only applies to patients who are discharged within this time period.
  For patients surviving to discharge and discharged within 14 days post-operatively. Categorical variable for which the options are 'transfer to another hospital', 'transfer to rehabilitation unit', 'usual place of residence' and 'absconded'. A surrogate measure of short term functional outcome.

CONTACTS AND LOCATIONS:
Overall Officials: David Clark, Principal Investigator — University of Cambridge; Peter Hutchinson, Principal Investigator — University of Cambridge; Alexis Joannides, Principal Investigator — University of Cambridge; Angelos Kolias, Principal Investigator — University of Cambridge
Locations (1):
- University of Cambridge, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
After publication of the main results, the pooled dataset will be available to all members of the GNOS collaboration for secondary analysis, after judgement and approval of each proposed analysis by the central study team.
Supporting Information: Study Protocol
Time Frame: After publication of the main results.